CLINICAL TRIAL: NCT01633645
Title: A Phase II, Open-Label Trial of Bortezomib (VELCADE®) in Combination With Gemcitabine and Cisplatin in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Bortezomib in Combination With Gemcitabine and Cisplatin in Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, Prof. V.Georgoulias, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-LUC-2006
Record Dates: First submitted 2012-03-13; First posted 2012-07-04 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Non Small Cell Lung Cancer; Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Bortezomib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade/GEM/CDDP (Experimental): Bortezomib / Gemcitabine / Cisplatin
  Interventions: Drug: Bortezomib; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Bortezomib — Velcade
  Other Names: VELCADE 1 mg/m2 on days 1 and 8, of a 21-days treatment cycle for a maximum of 8 cycles
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 on days 1 and 8 of a 21-days treatment cycle for a maximum of 8 cycles
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin 70 mg/m2 on day 1 of a 21-days treatment cycle for a maximum of 8 cycles
  Other Names: CDDP

SUMMARY:
The primary objective of this study is to establish the objective response rate (complete response + partial response) following treatment with VELCADE in combination with cisplatin plus gemcitabine in patients with locally advanced (Stage IIIb) or metastatic (stage IV non-small cell lung cancer (NSCLC) who have not received prior antineoplastic therapy for advanced disease

DETAILED DESCRIPTION:
By its mechanism of action i.e., inhibiting protein degradation, VELCADE targets a wide-range of pathways that are relevant to tumor progression and therapy resistance. Preclinical data in cell lines indicate anti-tumor activity in NSCLC. Preliminary work in vivo (animal models) suggests an enhanced anti-tumor effect in combination with cytotoxic agents commonly used in the treatment of lung cancer, including gemcitabine and CPT-11 and additive tumor growth delay when combined with cisplatin or paclitaxel.

Platinum- or non-platinum- based combinations including the newer agents represent the standard front-line treatment for patients with stage IIIB/IV NSCLC. However, despite the introduction of the newer agents, the efficacy of cytotoxic chemotherapy seems to have reached a plateau. The incorporation of molecularly targeted agents in NSCLC treatment is likely to improve the treatment outcomes. Recently, an initial Phase 2 of VELCADE in combination with gemcitabine/carboplatin in the first-line treatment of NSCLC was completed. A response rate of 21% with impressive progression-free survival and overall survival rates of 5 and 11 months, respectively, were reported.

Combining VELCADE with a currently approved standard regimen such as cisplatin/gemcitabine, may lead to a better response rate, TTP, and OS than chemotherapy alone. VELCADE combined with gemcitabine and cisplatin has been shown safe in a phase I trial in patients with advanced solid tumors. The maximum tolerated dose (MTD) of VELCADE was 1 mg/m2 on either a weekly or a biweekly schedule when combined with gemcitabine 1000 mg/m2 and cisplatin 70 mg/m2. Treatment was generally well tolerated with the weekly regimen of VELCADE being associated with less myelotoxicity. Plasma pharmacokinetic profiles of gemcitabine and cisplatin were not altered by VELCADE. Interestingly enough, among 27 patients with NSCLC an encouraging response rate of 37% and disease stabilization rate of 52% was recorded.

In this trial VELCADE alone will be administered on the first treatment cycle to examine molecular correlates of VELCADE activity. Subsequent cycles will include the combination of VELCADE with cisplatin plus gemcitabine.

Data from the phase I study of VELCADE plus cisplatin/gemcitabine contributed to the selection of the drug doses for patients that will be enrolled in the current study. Specifically, the doses employed are those identified as the MTD level of the phase I study.

The anti-tumor activity of the combination of VELCADE and cisplatin/gemcitabine in the first-line treatment of NSCLC will be tested in this study according to a Simon 2-stage optimal design.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 years of age or older.
* NSCLC histologically or cytologically confirmed.
* Locally advanced (Stage IIIB) or metastatic (Stage IV) NSCLC.
* No prior systemic anti-neoplastic therapy for Stage IIIB/IV NSCLC (one prior line is allowed if given as adjuvant or neo-adjuvant therapy).
* Measurable disease per RECIST criteria.
* ECOG performance status score of 0 - 1.
* Life expectancy greater than 3 months.
* Female patients must be postmenopausal (for at least 6 months), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and have a negative serum or urine β-human chorionic gonadotropin (hCG) pregnancy test at screening.
* Patients (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to and able to comply with the protocol requirements and participate in the study before any study-related procedure not part of normal medical care is conducted.
* Patients (or their legally acceptable representatives) must have signed an informed consent for testing indicating, that they agree to participate in the correlative marker part of the study.

Exclusion Criteria:

* Peripheral neuropathy of Grade 2 or greater intensity, as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE Version 3.0).
* Previous treatment with VELCADE.
* Prior systemic anti-neoplastic therapies for Stage IIIB/IV NSCLC except if as neoadjuvant therapy for Stage IIIB.
* Any prior systemic anti-neoplastic therapy for NSCLC (i.e., prior chemotherapy, radiation therapy, prior monoclonal antibodies or any investigational drug or any major surgery) within 4 weeks before enrollment.
* Significant weight loss (documented < 10% body weight in the 6 weeks before enrollment).
* Inadequate organ function at the screening visit as defined by the following laboratory values:

  * Platelet count ≤ 100 x 109/L
  * Hemoglobin ≤ 8.0 g/dL (80 g/L)
  * Absolute neutrophil count (ANC) ≤ 1.5 x 109/L
  * AST ≥ 3 times the upper limit of the normal range (upper normal limit) or > 5 times the upper normal limit for subjects with liver metastases
  * ALT ≥ 3 times ULN or > 5 times the upper normal limit for subjects with liver metastases (Calculated creatinine clearance ≥ 45 mL/min, Total bilirubin ≥ 1.5 times Upper normal limit)
* Myocardial infarction within 6 months before randomization or has New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Central nervous system metastasis or brain metastases unless patients have been subjected to local radiation therapy and are clinically stable. Brain computed tomography or magnetic resonance imaging is required in symptomatic patients to rule out brain metastases but is not required in asymptomatic patients.
* Serious medical condition (such as severe hepatic impairment, pericardial disease, acute diffuse infiltrative pulmonary disease, systemic infections etc) or psychiatric illness likely to interfere with participation in this study
* Other malignancy within the past 5 years. Exceptions for the following if treated and not active: basal cell or non-metastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or International Federation of Gynecology and Obstetrics Stage 1 carcinoma of the cervix.
* History of allergic reaction attributable to compounds containing boron or mannitol.
* Pregnant or breast-feeding.
* Currently enrolled in another clinical research study or has received an investigational agent for any reason within 4 weeks before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 9 weeks
  Participants will be evaluated for response to the study treatment after the first three treatment cycles (cycle repeated every 21 days) and then every two treatment cycles (completion of cycles 5, 7, 9 etc.) until documentation of disease progression.

SECONDARY OUTCOMES:
Progression free survival | 1 year
  Progression free survival will be calculated from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
Overall survival | 1 year
  Overall survival will be calculated from date of randomization until the date of death from any cause, assessed up to 36 months
Number of participants with adverse events | Participants will be followed for adverse events up to 24 weeks
  Participants will be followed for adverse events appearance until the end of treatment administration (seven treatment cycles repeated every 21 days plus two more cycles according to psysician's decision)plus 30 more days after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Heraklion; Sofia Aggelaki, MD, Principal Investigator — University Hospital of Heraklion
Locations (5):
- Greece (5):
  - Air Forces Military Hospital of Athens Athens, Greece, Athens
  - METAXA Hospital, B' Pathology Department, Athens
  - SOTIRIA Hospital, Medical Oncology Department, Athens
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki